CLINICAL TRIAL: NCT06970041
Title: To Assess the Types of Mechanical Ventilation in Enabling Therapeutic Bronchofiberoscopy in Patients With Decompensated Respiratory Acidosis (Complete Respiratory Failure)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BNW/NWN/0052/KB1/96/I/24/25
Record Dates: First submitted 2025-04-04; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Failure With Hypercapnia; Therapeutic Bronchofiberoscopy
Keywords: Bronchofiberoscopy (FOB); High Flow Nasal Cannula (HNFC); Non-Invasive Ventilation (NIV); Passive Oxygen Therapy; Type 2 respiratory failure; Exacerbation of Chronic Respiratory Acidosis; Invasive Mechanical Ventilation (IMV)
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- pH < 7,2, NIV (Active Comparator): The use of NIV in patients undergoing therapeutic FOB with the most severe type 2 respiratory failure
  Interventions: Device: Use of NIV during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure
- pH < 7,2, IMV (Intubation) (No Intervention): The use of IMV in patients undergoing therapeutic FOB with the most severe type 2 respiratory failure (current gold standard at ICU fascilities)
- 7,3> pH ≥ 7,2, NIV (Active Comparator): The use of NIV in patients with type 2 respiratory failure undergoing therapeutic FOB with a pH level: 7,3> pH ≥ 7,2.
  Interventions: Device: Use of NIV during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure
- 7,3> pH ≥ 7,2, HFNC (Active Comparator): The use of HFNC in patients with type 2 respiratory failure undergoing therapeutic FOB with a pH level: 7,3> pH ≥ 7,2.
  Interventions: Device: Use of HFNC during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure
- 7,35> pH ≥ 7,3, NIV (Active Comparator): The use of NIV in patients with type 2 respiratory failure undergoing therapeutic FOB with a pH level: 7,35> pH ≥ 7,3
  Interventions: Device: Use of NIV during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure
- 7,35> pH ≥ 7,3, HFNC (Active Comparator): The use of HFNC in patients with type 2 respiratory failure undergoing therapeutic FOB with a pH level: 7,35> pH ≥ 7,3
  Interventions: Device: Use of HFNC during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure
- 7,35> pH ≥ 7,3, Passive Oxygen Therapy (control group) (No Intervention): The use of passive oxygen therapy (current gold standard) in patients with type 2 respiratory failure undergoing therapeutic FOB with a pH level: 7,35> pH ≥ 7,3

INTERVENTIONS:
Device: Use of NIV during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure — The aim of the project is to assess the safety, indications and contraindications for therapeutic bronchofiberoscopy in patients with decompensated respiratory acidosis using: invasive mechanical ventilation (IMV), non-invasive mechanical ventilation (NIV) and high-flow nasal canulla (HFNC). Additionally, we want to determine to what extent the use of respiratory support during bronchofiberoscopy (BF) will avoid complications such as exacerbation of hypoxemia and/or acidosis and the occurrence of hemodynamic instability.
  Arms: 7,35> pH ≥ 7,3, NIV; 7,3> pH ≥ 7,2, NIV; pH < 7,2, NIV
Device: Use of HFNC during therapeutic FOB as a respiratory support method in patients with type 2 respiratory failure — The aim of the project is to assess the safety, indications and contraindications for therapeutic bronchofiberoscopy in patients with decompensated respiratory acidosis using: invasive mechanical ventilation (IMV), non-invasive mechanical ventilation (NIV) and high-flow nasal canulla (HFNC). Additionally, we want to determine to what extent the use of respiratory support during bronchofiberoscopy (BF) will avoid complications such as exacerbation of hypoxemia and/or acidosis and the occurrence of hemodynamic instability.
  Arms: 7,35> pH ≥ 7,3, HFNC; 7,3> pH ≥ 7,2, HFNC

SUMMARY:
Background:

Bronchofiberoscopy (FOB) is a minimally invasive and safe procedure performed for diagnostic and therapeutic purposes. FOB frequently impairs respiratory function, which may lead to possible exacerbation of respiratory failure.

Currently, the most frequent respiratory support is passive oxygen therapy, but non-invasive ventilation (NIV) and high flow nasal cannula (HFNC) are increasingly attempted, however the optimal setting and indications for NIV and HFNC in patients undergoing FOB with respiratory acidosis, haven't been determined yet.

Methods:

The study protocol describes a prospective, multicenter, three-armed randomized controlled trial (RCT).

The investigators aim to study patients undergoing a therapeutic bronchofiberoscopy with decompensated type 2 respiratory failure: (pH <7.35 and pCO2 >45 mmHg);

1. randomized to: passive oxygen, NIV, HFNC, invasive mechanical ventilation (IMV);
2. total number of participants: 315. Before FOB, the patient group will undergo arterial blood gas analysis (ABG). During FOB there will be a continuous monitoring of vital signs as in: SpO2, FiO2, TcCO2, ECG, and Heart Rate. After FOB, the investigators are going to perform another ABG, mark endpoints, and complications, if any arise.

Results:

Based on the selected endpoints, or any complication related to FOB the investigators hope to determine which of the respiratory methods: passive oxygen, NIV, HFNC or IMV provides the best support, leading to a lower number of complications and overall a better tolerance of FOB by the patient. Additionally, our aim is to find the optimal settings for NIV and HFNC in the studied group.

Conclusions:

The results of this study are going to assess the need and the role of the optimal respiratory support method among patients with exacerbation of respiratory acidosis, leading to a shorter time from admission to full recovery, better tolerance during the procedure, quicker recovery after procedure.

DETAILED DESCRIPTION:
To assess the types of mechanical ventilation in enabling therapeutic bronchofiberoscopy in patients with decompensated respiratory acidosis (complete respiratory failure).

The aim of the project The aim of the project is to assess the safety, indications and contraindications for therapeutic bronchofiberoscopy in patients with decompensated respiratory acidosis using: invasive mechanical ventilation, non-invasive mechanical ventilation (NIV) and high-flow nasal canulla (HFNC). Additionally, the investigators want to determine to what extent the use of respiratory support during bronchofiberoscopy (BF) will avoid complications such as exacerbation of hypoxemia and/or acidosis and the occurrence of hemodynamic instability.

Project justification

Bronchofiberoscopy is a safe procedure that has great therapeutic value for respiratory diseases. BF plays an important role in the diagnosis of hemoptysis, respiratory infections, interstitial lung diseases, lung tumors, mediastinal lymphadenopathy, and evaluation of transplanted lungs. bronchoscopy may have therapeutic applications in cases of foreign body aspiration and the need to perform bronchial toilet.

Regardless of the indications, airway narrowing occurs during BF, which may exacerbate respiratory failure and secondarily influence the occurrence of cardiac and pulmonary complications.

Sedation, which improves the tolerance of the procedure, may also lead to increased respiratory failure. For this reason, respiratory support methods are increasingly used in people with circulatory and respiratory burdens during the procedure. The basic technique of respiratory support is the use of standard nasal cannulas enabling passive oxygen therapy. Due to the increasing number of seriously ill patients with respiratory failure, passive oxygen therapy is often an insufficient method to safely perform BF. So far, most of these patients were disqualified from BF or intubation was required.

NIV prevents the collapse of peripheral airways, reduces the number and size of atelectasis foci and prevents their formation, and helps to treat hypercapnic respiratory failure. NIV, through the recruitment of pulmonary alveoli, leads to an increase in vital capacity and lung compliance, and also reduces the workload on the heart. NIV may enable therapeutic bronchofiberoscopy in patients with pulmonary alveolar proteinosis without the need for intubation. NIV enables safe performance of therapeutic bronchofiberoscopy in patients with exacerbation of respiratory failure and in patients with severe chronic respiratory failure.

HFNC is an innovative method of respiratory support that allows for obtaining a high flow in nasal cannulas, heating and humidifying the air, and precise setting of the necessary oxygen concentration in the respiratory mixture up to FiO2 values reaching 1.0 (100%). Such a high flow is associated with another significant advantage of this method - generating constant positive airway pressure (CPAP), which additionally supports the mechanics of breathing.

NIV and HFNC are used to increase the safety of BF in patients with respiratory failure. At present, there are no evidence-based data defining differences in the safety profile and indications justifying the choice of NIV-BF or HFNC-BF.

Moreover, no specific indications and contraindications for the above-mentioned procedures have been determined, as there are no prospective randomized studies to date that would indicate the superiority of one of the techniques in patients with respiratory acidosis.

Currently, there are no universal disease-specific settings for both devices that could be used during bronchoscopy in patients with acute respiratory acidosis, chronic respiratory acidosis or its exacerbations. In patients with severe respiratory failure, intubation should be considered before the procedure to enable safe bronchofiberoscopy. In patients who have not been intubated, bronchofiberoscopy may cause exacerbation of respiratory failure, which may lead to the need for urgent intubation, transfer to the ICU or sudden cardiac arrest in a patient undergoing bronchofiberoscopy.

Intubation of the patient further increases tracheal stenosis and prevents the insertion of a standard bronchoscope in the case of endotracheal tubes smaller than 7.5-8 mm in diameter.

The use of such a tube causes the degree of narrowing of the airways through which the patient is ventilated to be much greater, because between the bronchoscope and the endotracheal or tracheostomy tube, even in the case of a size of 8-8.5 mm, there is only a very narrow slit-like lumen outside the bronchoscope, which, drawing from the formula for flow resistance according to Poiseuille's law, generates an increase in resistance.

Therefore, intubating a patient for bronchofiberoscopy will require the use of very high ventilation pressures during the procedure, because in other cases the tidal volume will decrease and respiratory failure will increase. Generating these pressures creates a risk of complications such as barotrauma and decreased blood pressure. When deciding to intubate a patient, the widest possible endotracheal tube should be used, which increases the risk of vocal cord injury. Despite this, in order to provide ventilation during BF in an intubated patient, the narrowing of the airways encourages the use of a narrower bronchofiberscope. A narrower bronchofiberscope will have a smaller working channel, reducing the effectiveness of bronchofiberscopies performed especially for therapeutic indications.

The study will be conducted in departments dealing with patients with respiratory failure: in pulmonary departments; in bronchoscopic laboratories, where patients from various departments are treated, e.g. cardiology departments, internal medicine departments; in ICUs in patients who were not intubated a priori. The study is to assess the best and safest indications for performing BF depending on the severity and type of respiratory acidosis.

The subject of our study is particularly important because by defining the indications and criteria for the use of respiratory support in the form of NIB and HFNC during bronchofiberoscopy, it will be possible to perform this procedure in a larger group of patients who would initially be disqualified from this procedure. Additionally, it will reduce the group of patients who would require intubation for bronchofiberoscopy. Moreover, the use of HFNC or NIV may probably reduce the risk associated with BF and sedation.

Therefore, no new prospective studies were performed in this area, because it has been proven that intubation allows for the performance of BF in patients with complete respiratory failure.

Silesian Medical University Bioethics Committee (SUM BC) the protocol, Resolution No: BNW/NWN/0052/KB1/96/I/24/25

CPAP was not included in the randomization of the study groups because, although it improves oxygenation, it is not an acceptable ventilation mode. CPAP does not generate pressure support (PS), and ultimately the reduced work of breathing is caused by the recruitment of pulmonary alveoli. In addition, HFNC has the ability to generate positive end-expiratory pressure (PEEP) of up to about 5 cm3, with the mouth closed, which is significantly limited during BF. Additionally, most of the devices used recently in bronchoscopic laboratories have both modes of operation: NIV and CPAP, therefore it seems more reasonable to use NIV, which pathophysiologically should be more effective and safer in patients administered sedation.

Study group

The study will include patients (women and men) who express informed consent to participate in the proposed study. Recruitment will be conducted in people ≥18 years of age with indications for urgent bronchofiberoscopy.

A conversation will be conducted with patients in conditions of maintaining privacy and meeting the GDPR criteria. Patients will be thoroughly informed about the course of the study, encouraged to ask questions, with full explanation of doubts. Then, patients will be asked to provide written consent to participate in the research project.

The target planned number of 315 patients studied from all groups, 105 in each arm, which was calculated based on the risk of complications in the form of intubation during BF in patients with respiratory failure with a frequency estimated at 0.2-2%. In the group of the most seriously ill patients (pH < 7.2), after recruiting 15, 30, and 45 patients, respectively, a partial analysis will be performed to enable monitoring of the study safety in the group of patients at highest risk of complications.

Research methodology The protocol assumes the launch of a multicenter, international prospective randomized trial (RCT). Patients will be assigned to each of the study arms based on the pH level in blood gasometry. In each arm, patients will be randomly assigned to one of two dedicated methods of respiratory support (Figure. 2: Randomization).

The last prospective data on patients with complete respiratory failure requiring BF come from the 1970s, where it was proven that intubation of the patient enables this examination to be performed.

A detailed medical history will be collected from the patients (including comorbidities, medications taken, smoking history and NYHA, mMRC, Charslon scale, CCS, BORG, Apache II, SAPS II, RASS questionnaires). Blood pressure, saturation will be measured and a blood gas (approximately 2.0 ml) will be taken to classify the patient into one of the three groups (Figure 1 and 2). Blood gas analysis before the examination will have to be performed in such a way as to enable precise determination of pCO2, pH and HCO-3 (given FiO2 and type of respiratory support used). After the patient has been classified into a specific section, they will be randomly assigned to a given method of respiratory support during the bronchoscopic examination.

Course of the study and escalation of therapy In the case of high-flow oxygen therapy, the patient will be fitted with special nasal cannulas and then an examination will be performed. In the case of NIV, the patient will be fitted with a non-invasive ventilation mask with a special bronchoscopic elbow containing a valve enabling the introduction of a bronchofiberscope. The study will compare the initial settings of the devices, which will be maintained provided that the examination is carried out correctly and the patient's clinical condition is stable. In the case of desaturations, hypercapnia or other abnormalities in the assessment of the patient, the settings may be changed or the method may be converted based on the principle of therapy escalation (HFNC → NIV →MV).

Monitoring During the entire examination, parameters such as SpO2, FiO2, TcCO2, ECG and heart rate (these parameters will be monitored continuously) as well as arterial blood pressure using a non-invasive method (measured every 5 minutes) will be monitored.

After BF

After bronchofiberoscopy, blood gas analysis will be repeated and endpoints and complications such as bronchospasm, hypoxemia, decompensated respiratory acidosis, local bleeding, fever, need to interrupt the procedure, transfer to the ICU, pneumothorax, death will be recorded. BF will be performed using optical or video bronchofiberscopes or endobronchial endosonography (EBUS) devices. The diameter of the bronchofiberscope used should be recorded as well as the type and dose of sedation used during BF in each of the three randomized groups, however, bearing in mind that the depth of sedation should be within the RASS range of -2 to -3.

Data obtained from the interview and additional tests will be anonymously entered into a computer database in compliance with GDPR criteria and then statistically processed. Appropriate conclusions will be drawn based on the results obtained.

Randomization Randomization will be performed. The database and online randomization platform will be assessable for participating centers online at www.pneumosilesia.org available for collaborating centers after receiving their BC approval.

The patients undergoing FOB for therapeutic reasons will be randomized after being assigned to a subgroup previously mentioned based on their pH level. After categorizing them, in each group there will be a randomization for the specific respiratory support method.

1. Therapeutic FOB , randomization within shown groups:

a. pH< 7.2 (105 patients) i. MV ii. NIV b. 7.2 ≤ pH < 7.3 (105 patients) i. NIV ii. HFNC c. 7.3 ≤ pH < 7.35 (105 patients) i. NIV ii. HFNC iii. Passive oxygen therapy

Device setting

1. HFNC, flow 60L/min, temperature 34oC and FiO2 under saturation control to achieve SpO2≥92% Baseline FiO2 - equivalent to FiO2 during oxygen therapy before BF (during hospitalization),
2. NIV will be conducted in ST mode (spontaneous to forced), number of breaths 16-18/minute, EPAP (positive expiratory pressure) 6-14 cmH2O, Tins (duration) 0.8-1s, PS 8-25 cm H2O and oxygen flow under saturation control to achieve SpO2≥92% (baseline oxygen with FiO2 - at the level of previously administered FiO2, trigger and low cycle
3. MV: device parameters will correspond to previous settings to achieve SpO2≥92%, based on minute ventilation and tidal volume. The initial mode used should be recorded, including PS, EPAP, and FiO2. For intubated patients, the endotracheal tube size should be recorded.

Project duration: 3 years Partner centres will be obliged to apply to their relevant bioethics committees and to cover their patients with appropriate insurance.

Expected Endpoints

* Possibility of performing bronchoscopy (therapeutic) in patients who were initially disqualified,
* Improved patient comfort during the examination, thanks to the use of deeper sedation,
* Increased safety and comfort of BF in patients with respiratory failure (decrease in the number of procedures in which mild and severe complications occurred)
* Endpoints and complications such as prolonged hospitalization, bronchospasm, hypoxemia episode, decompensated respiratory acidosis, local bleeding, fever, need to interrupt the procedure, transfer to the ICU, pneumothorax, death will be marked.

Funding:

The work was supported by the Silesian Medical University (BNW-1-118/N/4/K).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age with indications for bronchoscopy:

   Therapeutic examination: pneumonia in people with impaired cough reflex, culture and toilet of the bronchial tree, respiratory tract hemorrhages treated with a bronchofiberoscope and aspiration of a foreign body, bronchial unblocking in advanced neoplastic disease.
2. Patient who signed a written informed consent to participate in the study,
3. pCO2 > 45 mmHg and pH < 7.35 in a blood gas analysis performed directly during qualification for FOB.

Exclusion Criteria:

1. Lack of written, informed consent of the subject to participate in the research project,
2. Unstable coronary artery disease chronic coronary syndrome (CCS) III/IV, circulatory failure New York Heart Association (NYHA) III/IV (does not apply to tests for vital indications, e.g. aspiration of a foreign body),
3. Hemodynamic insufficiency, constant use of pressor amines, myocardial infarction in the last 2 weeks without percutaneous coronary intervention (PCI) treatment, unstable angina pectoris, severe arrhythmias- especially ventricular,
4. Chronic primary pulmonary hypertension, assessed during right heart catheterization WHO III/IV,
5. Pneumothorax not secured with drainage,
6. Platelet count <20,000/µl, if platelets are not transfused immediately before or during the procedure,
7. International normalized ratio (INR)> 2 or activated partial thromboplastin time (APTT) > 36 s, in the case of therapeutic FOB [16],

d. Anemia: hemoglobin (Hb) level <6 g/dl or 6-10 g/dl if the physician prescribes a blood transfusion, h. Patients who were intubated before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
NIV allows for a safe therapeutic bronchoscopy in patients with type 2 respiratory failure. | During the procedure, and after up to the arterial blood gas analysis (1day)
  The investiagators are going to asses the performance of NIV in patients with type 2 respiratory failure undergoing a therapeutic FOB marking endpoints such as:
  * Hypoxemia, decrease in saturation >5% for more than 30 seconds,
  * PO2 before and after FOB from blood gas analysis,
  * PO2/FiO2 before and after FOB from blood gas analysis,
  * Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study,
  * PCO2 before and after FOB from blood gas analysis,
  * pH before and after FOB from blood gas analysis,
  * Need to extend NIV therapy after FOB - [time in minutes],
  * Need to escalate NIV therapy, NIV -> intubation,
HFNC allows for a safe therapeutic bronchoscopy in patients with type 2 respiratory failure. | During the procedure, and after up to the arterial blood gas analysis (1day)
  The investiagators are going to asses the performance of HFNC in patients with type 2 respiratory failure undergoing a therapeutic FOB marking endpoints such as:
  * Hypoxemia, decrease in saturation >5% for more than 30 seconds,
  * PO2 before and after FOB from blood gas analysis,
  * PO2/FiO2 before and after FOB from blood gas analysis,
  * Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study,
  * PCO2 before and after FOB from blood gas analysis,
  * pH before and after FOB from blood gas analysis,
  * Need to extend HFNC therapy after FOB - [time in minutes],
  * Need to escalate HFNC therapy, HFNC-> NIV; NIV -> intubation,
The number of complications after a therapeutic FOB in patients with type 2 respiratory failure | Through study completion, an average of 1 years
  Endpoints and complications such as prolonged hospitalization, bronchospasm, hypoxemia episode, decompensated respiratory acidosis, local bleeding, fever, need to interrupt the procedure, transfer to the ICU, pneumothorax, death will be marked.

SECONDARY OUTCOMES:
HFNC device setting for patients with type 2 respiratory failure undergoing bronchoscopic procedures | During the procedure, and after up to the arterial blood gas analysis (1day)
  For therapeutic FOB the HFNC setting will be set to:
  HFNC, flow 60L/min, temperature 34oC and FiO2 under saturation control to achieve SpO2≥92% Baseline FiO2 - equivalent to FiO2 during oxygen therapy before FOB (during hospitalization),
  During FOB all needed changes in settings for a safe procedures will be marked, by measurment of parameters for the optimal setting choice:
  Hypoxemia, decrease in saturation >5% for more than 30 seconds, PO2 before and after FOB from blood gas analysis, PO2/FiO2 before and after FOB from blood gas analysis, Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study, PCO2 before and after FOB from blood gas analysis.
NIV device setting for patients with type 2 respiratory failure undergoing bronchoscopic procedures | During the procedure, and after up to the arterial blood gas analysis (1day)
  For therapeutic FOB the NIV setting will be set to:
  NIV will be conducted in ST mode (spontaneous to forced), number of breaths 16-18/minute, EPAP (positive expiratory pressure) 6-14 cmH2O, Tins (duration) 0.8-1s, PS (pressure support ventilation) 8-25 cm H2O and oxygen flow under saturation control to achieve SpO2≥92% (baseline oxygen with FiO2 - at the level of previously administered FiO2, trigger and low cycle
  During FOB all needed changes in settings for a safe procedures will be marked, by measurment of parameters for the optimal setting choice:
  Hypoxemia, decrease in saturation >5% for more than 30 seconds, PO2 before and after FOB from blood gas analysis, PO2/FiO2 before and after FOB from blood gas analysis, Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study, PCO2 before and after FOB from blood gas analysis.
MV device setting for patients with type 2 respiratory failure undergoing bronchoscopic procedures | During the procedure, and after up to the arterial blood gas analysis (1day)
  For therapeutic FOB the MV setting will be set to:
  MV: device parameters will correspond to previous settings to achieve SpO2≥92%, based on minute ventilation and tidal volume. The initial mode used should be recorded, including PS, EPAP, and FiO2. For intubated patients, the endotracheal tube size should be recorded.
  During FOB all needed changes in settings for a safe procedures will be marked, by measurment of parameters for the optimal setting choice:
  Hypoxemia, decrease in saturation >5% for more than 30 seconds, PO2 before and after FOB from blood gas analysis, PO2/FiO2 before and after FOB from blood gas analysis, Hypercapnia measured transcutaneous TcCO2, increase in PCO2 >10 mm Hg for more than 30 seconds during the study, PCO2 before and after FOB from blood gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Szymon Skoczyński, PhD, professor of university, Principal Investigator — Department of Lung Diseases and Tuberculosis, Faculty of Medical Sciences in Zabrze, Medical University of Silesia, Katowice, Poland.